CLINICAL TRIAL: NCT00058773
Title: Administration of Autologous Neomycin Resistant Gene Marked EBV Specific Cytotoxic T-Lymphocytes as Therapy for Patients Receiving Autologous Bone Marrow Transplant for Relapsed EBV-Positive Lymphoma.
Brief Title: Giving Gene Marked EBV Specific T-Cells to Patients Receiving a BMT for Relapsed EBV-Positive Hodgkin Disease
Acronym: ANGELA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, catherine bollard, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-6422-ANGELA; ANGELA
Record Dates: First submitted 2003-04-11; First posted 2003-04-15 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Hodgkin Disease; Non-Hodgkins Lymphoma
Keywords: Hodgkin disease; non-Hodgkins Lymphoma; bone marrow transplant
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CTL Administration (Experimental): Infusion of EBV Specific Cytotoxic T-Lymphocytes
  Interventions: Drug: Infusion of EBV Specific Cytotoxic T-Lymphocytes

INTERVENTIONS:
Drug: Infusion of EBV Specific Cytotoxic T-Lymphocytes — EBV specific cytotoxic T-lymphocytes will be given by intravenous injection over 1-10 minutes.
  Each patient will receive two injections, 14 days apart.

SUMMARY:
Subjects have a type of lymph gland cancer called Hodgkin or non-Hodgkin Lymphoma, which has come back or not gone away after treatment, including the best treatment we know for relapsed Lymphoma. We are asking subjects to volunteer to be in a research study using Epstein Barr virus (EBV) specific cytotoxic T lymphocytes, a new experimental therapy. This therapy has never been used in patients with Hodgkin disease or this type of non-Hodgkin Lymphoma but it has been used successfully in children with other types of blood cancer caused by EBV after bone marrow transplantation.

Some patients with Hodgkin disease or non-Hodgkin Lymphoma show evidence of infection with the virus that causes infectious mononucleosis Epstein Barr virus (EBV) before or at the time of their diagnosis of Lymphoma. EBV is often found in the cancer cells suggesting that it may play a role in causing Lymphoma. The cancer cells infected by EBV are very clever because they are able to hide from the body's immune system and escape destruction. We want to see if we can grow special white blood cells, called T cells, that have been trained to kill EBV infected cells and give them back to subjects.

DETAILED DESCRIPTION:
We will take 60-70 ml (12 teaspoonfuls) of blood from the subject. We will first make a B cell line called a lymphoblastoid cell line or LCL by infecting the subjects blood with a laboratory strain of EBV called B95. We will then use use this EBV infected cell line (which have been treated with radiation so that they cannot grow) as stimulator cells and mix it with more blood. This stimulation will train the T cells to kill EBV infected cells and result in the growth of an EBV specific T cell line. We will then test the T cells to make sure that they kill the EBV infected cells and not your normal cells and freeze them.

The cells will be thawed and injected into subjects over 10 minutes, after pretreatment with Tylenol and Benadryl. A total of two doses will be given two weeks apart. All of the treatments will be given at Texas Children's Hospital or The Methodist Hospital.

We will follow subjects in the clinic after the injections. At each visit about 10ml (2 teaspoonfuls) of blood will be taken every other week for 6 weeks after the injection and then every 3 months for 1 year to monitor the subjects blood chemistry and hematology.

To learn more about the way the T cells are working in the subjects body, an extra 40mls (8 teaspoons) of blood will be taken pre-infusion, 3-4 days post infusion (optional) and at 1, 2, 4 and 6 weeks post-infusion and then at 3, 6, 9, and 12 months. The blood may be drawn from the subjects central line at the time of their regular blood tests.

ELIGIBILITY:
INCLUSION CRITERIA:

* Any patient with Hodgkin disease or non-Hodgkin Lymphoma, containing the EBV genome or antigen, receiving an autologous bone marrow transplant regardless of age or sex.
* Patients with tumor tissue EBV +ve.
* Patients with life expectancy >6 weeks.
* Patients with Karnofsky score of > 50.
* No severe intercurrent infection.
* Patient, parent/guardian able to give informed consent.
* Patient with Bilirubin <2x normal, SGOT <3x normal, and ANC greater than 500mm
* Patients with creatinine <2x normal for age or creatinine clearance >2x normal for age.
* Patients should have been off other investigational therapy for one month prior to entry in this study.

EXCLUSION CRITERIA:

* Patients with a life expectancy of <6 weeks.
* Patients with an EBV positive Lymphoma secondary to an acquired or congenital immunodeficiency.
* Patients with a Karnofsky score less than or equal to 50.
* Patients with a severe intercurrent infection.
* Patients with a bilirubin >2x normal,SGOT >3x normal, or abnormal prothrombin time.
* Patients with a creatinine >2x normal for age or creatinine clearance <2x normal for age.
* Patients with an ANC <500mm
* Patient, parent/guardian unable to give informed consent.
* Patients who have been on other investigational therapy within one month prior to entry in this study.
* Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. Women of childbearing potential must be on appropriate birth control for the duration of the study and 6 months after completion of the study. In addition, the male partner should use a condom.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1996-01; Primary Completion 2002-04 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
determine the safety of 2 IV injections of autologously derived EBV specific cytotoxic T-lymphocytes | 8 weeks
  The two injections will be given at day 0 and day 14. Three patients will be enrolled at the first dose level and followed for six weeks after the second dose (which will constitute a course) for evaluation of any critical toxicity.

SECONDARY OUTCOMES:
determine the survival, immunological efficacy and anti-tumor effects of EBV specific cytotoxic T-lymphocyte lines. | 1 year
  During the course of the study the survival, immunological efficacy and anti-tumor activity of neomycin resistance gene marked EBV specific cytotoxic T-lymphocyte lines will also be studied. In order to get a reasonable insight into the anti-tumor activity and late toxicity the patients will be followed for additional six weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bollard, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas